CLINICAL TRIAL: NCT05409157
Title: A Phase 1, Single-center, Open-label Study to Evaluate the Pharmacokinetics, Metabolism, and Excretion of [14C] BMS-986166 in Healthy Male Participants
Brief Title: A Study to Evaluate the Drug Levels of BMS-986166 in Healthy Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IM018-010
Record Dates: First submitted 2022-06-03; First posted 2022-06-08 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Healthy Participants
MeSH Terms: interventions — BMS-986166; Bisacodyl

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment Group 1: BMS-986166 (Experimental)
  Interventions: Drug: BMS-986166; Drug: Bisacodyl

INTERVENTIONS:
Drug: BMS-986166 — Specified dose on specified days
Drug: Bisacodyl — Specified dose on specified days
  Other Names: Dulcolax®

SUMMARY:
The purpose of this study is to assess the drug levels of BMS-986166 in healthy male participants.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male participants as determined by no clinically significant deviation from normal in medical history, physical examination, 12-lead ECGs, or clinical laboratory determinations
* Body mass index between 18.0 to 33.0 kg/m2 (inclusive)

Exclusion Criteria:

* Any significant acute or chronic medical illness
* Current or recent history of constipation or irregular bowel movement (less than 1 bowel movement per day within the last 1 week)
* History of allergy (such as rash, hives, breathing difficulties) to any medications, either prescription or nonprescription

Other protocol-defined inclusion/exclusion criteria apply

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2022-06-17 (Actual); Primary Completion 2022-10-15 (Actual); Study Completion 2022-10-15 (Actual)

PRIMARY OUTCOMES:
Total amount of total radioactivity (TRA) recovered in urine (UR) | Up to 90 days
Total amount of TRA recovered in feces (FR) | Up to 90 days
Total amount of TRA recovered in urine and feces combined (RTotal) | Up to 90 days
Percent of TRA recovered in urine (%UR) | Up to 90 days
Percent of TRA recovered in feces (%FR) | Up to 90 days
Percent of TRA recovered in urine and feces combined (%TOTAL) | Up to 90 days
Maximum observed concentration (Cmax) | Up to 89 days
Time of maximum observed concentration (Tmax) | Up to 89 days
Area under the concentration-time curve from time zero to time of the last quantifiable concentration [AUC(0-T)] | Up to 89 days

SECONDARY OUTCOMES:
Number of participants with adverse events (AEs) | Up to 124 days
Number of participants with serious adverse events (SAEs) | Up to 124 days
Number of participants with vital sign abnormalities | Up to 90 days
Number of participants with electrocardiogram (ECG) abnormalities | Up to 90 days
Number of participants with physical examination abnormalities | Up to 90 days
Number of participants with clinical laboratory test abnormalities | Up to 90 days
Maximum observed concentration (Cmax) | Up to 89 days
Time of maximum observed concentration (Tmax) | Up to 89 days
Area under the concentration-time curve from time zero to time of the last quantifiable concentration [AUC(0-T)] | Up to 89 days

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution - 0001, Madison, Wisconsin, United States

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome